CLINICAL TRIAL: NCT00346957
Title: A Phase II Study of Anecortave Acetate for the Treatment of Exudative Age-Related Macular Degeneration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-98-03
Record Dates: First submitted 2006-06-28; First posted 2006-07-04 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: AMD
MeSH Terms: interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Anecortave Acetate 30 (Experimental)
  Interventions: Drug: Anecortave acetate 30 mg
- Anecortave Acetate 15 (Experimental)
  Interventions: Drug: Anecortave Acetate 15 mg
- Anecortave Acetate 3 (Experimental)
  Interventions: Drug: Anecortave Acetate 3 mg
- Anecortave Acetate Vehicle (Placebo Comparator)
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave acetate 30 mg — 0.5ml administered onto the sclera once every six months for 24 months
  Arms: Anecortave Acetate 30
Drug: Anecortave Acetate 15 mg — 0.5ml administered onto the sclera once every six months for 24 months
  Arms: Anecortave Acetate 15
Drug: Anecortave Acetate 3 mg — 0.5ml administered onto the sclera once every six months for 24 months
  Arms: Anecortave Acetate 3
Other: Anecortave Acetate Vehicle — 0.5ml administered onto the sclera once every six months for 24 months
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of the study is to determine the concentration of anecortave acetate (15 or 30 mg versus placebo) that is safe and effective for the inhibition of the growth of blood vessels in the retina in patients with wet AMD.

ELIGIBILITY:
Inclusion Criteria:

* Ages 50 years and over
* Other protocol-defined inclusion and exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 1999-04; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Mean change in logMAR visual acuity at 12 months from baseline. | 12 months